CLINICAL TRIAL: NCT04638972
Title: An In-Vivo Evaluation of the Accuracy of Different Generation Apex Locators and Tactile Sense in Primary Teeth
Brief Title: Accuracy of Apex Locators in Primary Teeth
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Seçil Çalışkan, Assistant Professor, Eskisehir Osmangazi University
Other Study IDs: E25403353-050.99-107474
Record Dates: First submitted 2020-11-12; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Endodontically Treated Teeth; Primary Teeth; Pulp Necroses
MeSH Terms: conditions — Tooth, Nonvital; Dental Pulp Necrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Tactile Sense Method: In clinical practice, tactile sense and conventional radiography have been the methods of choice for determination of working length for a long time. However, these two methods have some limitations in determining working length. While the accuracy rate in tactile sense changes with experience, radiographic examination in children is usually hard due to poor cooperation or the unsuitable sensor size for child's small mouth [7]. Also, these techniques may yield inaccurate information especially in cases with root resorption
  Interventions: Device: working length determination techniques
- Radiographic Method (digital periapical radiography): In clinical practice, tactile sense and conventional radiography have been the methods of choice for determination of working length for a long time. However, these two methods have some limitations in determining working length. While the accuracy rate in tactile sense changes with experience, radiographic examination in children is usually hard due to poor cooperation or the unsuitable sensor size for child's small mouth [7]. Also, these techniques may yield inaccurate information especially in cases with root resorption
  Interventions: Device: working length determination techniques
- Ipex® EAL: Electronic apex locaters (EALs), which are based on electrical principles instead of visual determinants, have been used more frequently in primary teeth.
  Interventions: Device: working length determination techniques
- Propex® pixi EAL: Electronic apex locaters (EALs), which are based on electrical principles instead of visual determinants, have been used more frequently in primary teeth.
  Interventions: Device: working length determination techniques

INTERVENTIONS:
Device: working length determination techniques — A total of 30 infected mandibular primary second molar teeth in twelve children aged between 5 and 8 years were included in this study. Working length determination was performed using tactile sense, radiographic method and two different varieties of electronic apex locators (ProPex Pixi® and Ipex®) separately.

SUMMARY:
The aim of this study was to evaluate the effectiveness of tactile sense, digital periapical radiograph and two different varieties of electronic apex locators at working length determination in primary molars.

A total of 30 infected mandibular primary second molar teeth in twelve children aged between 5 and 8 years were included in this study. Working length determination was performed using tactile sense, radiographic method and two different varieties of electronic apex locators (ProPex Pixi® and Ipex®) separately.

DETAILED DESCRIPTION:
The teeth were first anaesthetized with Ultracaine Ds-Forte (Sanofi Aventis, İstanbul, Türkiye) and then isolated with rubber dam. Caries was removed and access cavity was prepared using a round diamond bur with copious water in each tooth. Barbed broaches were used to extirpate the pulpal tissue and 2.5 % sodium hypochlorite was used as the irrigation solution. Sterile cotton pellets were used to dry the cavity.

For working length determination, the groups were performed as; Group 1: Tactile Sense Method Group 2: Radiographic Method (digital periapical radiography) Group 3: Ipex® EAL Group 4: Propex® pixi EAL The measurement techniques given in the groups were used in each root canal of all primary molars (n=90).

Root canal length determination by tactile sense method:

In the determination of working length using tactile sense, a K-file with the tip that best adjusted to the apical area was selected and gently inserted into the canal until the operator felt the narrowest region. The silicone stop was then placed at the coronal reference, and tooth length considering the end of the root was measured with an endodontic ruler (0.5mm accuracy).

Root canal length determination by radiographic method:

In group 2, working length determination was performed with digital periapical radiograph (……………….). Before the radiographic evaluation, the protective thyroid lead and protective lead apron were used for all children. Digital periapical radiograph was taken with using paralleling technique while the files were in the canals. X-ray positioning device (FPS 3000-Film positioning system complete, TPC Advanced Technology Inc., California, USA) was used to standardize the distances between the source and the tooth, and the tooth and the film. Cusp adjacent to the canal was taken as the occlusal reference. Files, 1 mm shorter than the tooth length as recorded according to the preoperative radiograph, were inserted in the canals. The difference between the tip of the file and the end of the root was calculated on the image. In case the file had not passed the apex, this amount and the original length was calculated. In case the file had passed the apex, the amount was subtracted from the original length. Lastly, 1 mm was subtracted from this adjusted length to confirm the cemento-dentinal junction and recorded as radiographic working length.

Root canal length determination by EALs:

The electronic working length determination was performed either with Ipex®/Goup 2 (NSK Ltd, Tokyo, Japan) or ProPex Pixi®/Group 3 (Dentsply Maillefer, Ballaigues, Switzerland) apex locators. Lip clip was attached to patients' lower lip in order to complete the circuit. Then, the root canals were moistened with 0.9% saline solution, and a no.15 K- file (Dentsply Maillefer, Baillaigues, Switzerland) mounted to the holder was gently inserted till "0.5" signaled on the screen, meaning that the tip of file was at the apical constriction. If the reading was stable for at least 5 seconds, the file was pulled back and the length between the silicone stopper and the tip of the file was measured with an endodontic ruler.

Endodontic treatment was completed in same appointments.

ELIGIBILITY:
Inclusion Criteria:

- Children without any systemic diseases

Exclusion Criteria:

* Children with any systemic diseases as a contraindication to endodontic treatment (such as cardiac diseases, epilepsy etc.)
* Teeth with previous root canal manipulation, radiographic evidence of calcification, perforated pulpal floor, excessive internal root resorption, external resorption more than two-thirds of the root, excessive bone loss in the furcation and insufficient structure for restoration.

Ages: 5 Years to 8 Years | Sex: All
Age Groups: Child
Study Population: A total of 30 infected mandibular primary second molar teeth (90 canals) of twelve children aged between 5 and 8 years were included in this in vivo study
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Determination of root canal working length | 1 month
  Data were collected from measurements taken from each primary molar's root canal working length.
  Group 1: Tactile Sense Method Group 2: Radiographic Method (digital periapical radiography) Group 3: Ipex® EAL Group 4: Propex® pixi EAL The measurement techniques given in the groups were used in each root canal of all primary molars. After collection of the data, measurements taken from each root canal measurement method were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Seçil Çalışkan, Principal Investigator — Eskişehir Osmangazi University
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided